CLINICAL TRIAL: NCT04363307
Title: Prospective Study to Validate Ablation Parameters with MRI Based Scar for Left Atrial Ablation
Status: Completed | Type: Observational
Sponsor: Ravi Ranjan (Other)
Collaborators: Biosense Webster, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ravi Ranjan, Associate Professor, Cardiology, University of Utah
Organization: University of Utah (Other)
Other Study IDs: IRB_00130480
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adult participants: Adult participants ages 18 and older with AF
  Interventions: Device: AF Ablation; Device: MRI

INTERVENTIONS:
Device: AF Ablation — Adult participants undergoing standard of care AF ablation using VISITAG SURPOINT
Device: MRI — Adult participants will undergo a late gadolinium enhancement MRI of the left atrium three months post standard of care ablation

SUMMARY:
One of the goals of an ablation procedure is to create scarring of cardiac tissue. Not all ablations result in scar tissue. Advances in technology have improved scarring but ideal parameters that result in scar tissue are still not completely clear and there is great variability in the parameters used. Theoretically, intense ablation can always create scar tissue but is also likely to create more complications such as cardiac perforations. The investigator recently published another retrospective study looking at ablation parameters that reliably result in scar tissue but it had its limitations as it was retrospectively done.

This is a prospective study to validate the parameters that result in long term scarring. MRI has long been used to visualize ablation scar tissue. So in this study patients undergoing, initial left atrial ablation for atrial fibrillation as standard of care will undergo a 3 month post ablation MRI and that will be used to validate the ablation parameters.

DETAILED DESCRIPTION:
A critical step to improve atrial fibrillation (AF) ablation broadly is to minimize interoperator variability. VISITAG SURPOINT calculated a marker tag index value by combining contact force, power setting, and duration of energy delivered. Use of VISITAG SURPOINT has accurately predicted sites of pulmonary vein reconnection and regional changes in late gadolinium enhancement (LGE) and T2 (edema) intensity 24 hours post ablation. Prospective use of the ablation index improves first pass pulmonary vein isolation and 1-year freedom from atrial tachyarrhythmias compared to conventional treatment.

There remains a paucity of data regarding if ablation guided by index values and VISITAG SURPOINT results in durable scar formation in humans in general and compared to conventional approaches. In addition, the relative contribution of the components of VISITAG SURPOINT impact scar formation in-vivo and across a broad diversity of atrial anatomies. Such data are critical in patients that present with various degrees of atrial myopathies, arrhythmia substrate, and anatomies.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or early Persistent AF (continuous AF duration less than 3 months and CHADSVASC great than or equal to 2).
* First time ablation for AF
* Agreeable to a 3 month MRI

Exclusion Criteria:

* Claustrophobic (unable to undergo MRI)
* Having undergone prior left atrial ablation including AT or atypical flutter
* Metal implants that preclude getting an MRI
* eGFR < 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants ages 18 or older with paroxysmal or early persistent AF who will undergo their first ablation.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2020-05-14 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Correlation of ablative force with scar formation, on a scale of 0 (no correlation) to 1 (total correlation) | 3 months
Correlation of ablative power with scar formation, on a scale of 0 (no correlation) to 1 (total correlation) | 3 months
Correlation of ablation time on scar formation, on a scale of 0 (no correlation) to 1 (total correlation) | 3 months

SECONDARY OUTCOMES:
Change in circumferential extent of the lesion around pulmonary veins after ablation as measured by scar area | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Ranjan, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Health Sciences Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No